CLINICAL TRIAL: NCT06082466
Title: FRAMED Infrainguinal Venous Bypass Versus Conventional Autologous Bypass Trial
Acronym: Framed IVB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Klaus Linni, Head of Division of Vascular and Endovascular Surgery, MD PD, Paracelsus Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1144/2022
Record Dates: First submitted 2023-09-04; First posted 2023-10-13 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Occlusive Disease; Femoropopliteal Artery Occlusion; Femoropopliteal Stenosis; Critical Limb-Threatening Ischemia; Claudication, Intermittent
Keywords: Extraluminal Bypass Stenting; Autologous Vein Graft; Bypass Extremity Graft
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Autologous Bypass (Active Comparator)
  Interventions: Procedure: Conventional Autologous Bypass
- FRAMED Infrainguinal Venous Bypass (Active Comparator)
  Interventions: Procedure: FRAMED Infrainguinal Venous Bypass

INTERVENTIONS:
Procedure: FRAMED Infrainguinal Venous Bypass — The harvested vein graft will be covered with a mesh.
  Arms: FRAMED Infrainguinal Venous Bypass
Procedure: Conventional Autologous Bypass — The harvested vein graft will be used without a mesh coating.
  Arms: Conventional Autologous Bypass

SUMMARY:
The purpose of this clinical trial is to analyze patency after autologous infrainguinal bypass surgery in patients receiving a venous conduit versus a covered venous conduit.

DETAILED DESCRIPTION:
Patients presenting to Vascular Surgical Units are usually multimorbid with increased cardiopulmonary risk. Autologous venous bypass is indicated in certain situations despite the longer duration of surgery. Optimizing patency has been an important goal since many years. Reconstruction problems are often based on intimal hyperplasia, which can be reduced via covering of the harvested vein as seen in previous studies.

This clinical trial will be conducted at our Division of Vascular Surgery and Endovascular Surgery at the University Hospital of Salzburg. Patients will be randomized into one of the two treatment options, which are a plain venous conduit or a by mesh covered venous conduit. During this clinical trial, the first follow-up will take place after 6 weeks; this corresponds to the usual follow-up interval. Due to the trial, further follow-ups will take place for each of the patients after 3 months, 6 months, 12 months, 2 years.

ELIGIBILITY:
Inclusion Criteria

* Age at least 18 years
* Informed consent form with signature
* Rutherford Category 3 (<200m) or chronic critical ischemia (Rutherford Category 4-6)
* Assured inflow and recipient artery.

Exclusion Criteria

* Pregnant or breastfeeding women
* Active infection or sepsis
* Acute ischemia
* Endovascular procedure in the region to be treated.
* Vein with outer diameter <3.5 mm or >8 mm under pressure.
* Spliced Veins.
* Known allergy to the cobalt-chromium alloy (ASTM 1058) or its components (Cobalt-Chromium-Iron-Nickel-Molybdenum).
* Vasculitis
* Coagulopathy
* Radiation therapy near the anastomosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of primary patency of the venous bypass | 2 years
  The incidence of patency of the venous bypasses will be analysed and compared. This is defined as freedom from occlusion of the venous bypass.

SECONDARY OUTCOMES:
Incidence of procedure-related mortality | 2 years
  Mortality intervention-related
Incidence of 30-day mortality | 30 days
  Number of participants, who die within 30 days after the procedure.
Incidence of limb salvage after procedure | 2 years
  Amputation free survival

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Koter, MD, PD, Principal Investigator — Senior Physician; Stephanie Rassam, MD, Study Director — Resident Physician; Klaus Linni, MD, PD, FEBVS, Principal Investigator — Head of Division
Locations (1):
- University Hospital of Salzburg, Paracelsus Medical University, Salzburg, Austria